CLINICAL TRIAL: NCT03488563
Title: A Prospective, Randomized, Vehicle-Controlled, Double-Blind, Phase 2 Study to Assess the Safety, Tolerability, and Efficacy of B244 Delivered as an Intranasal Spray for Preventive Treatment in Subjects With Episodic Migraine
Brief Title: Study to Determine Safety and Efficacy of B244 in Subjects With Episodic Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AOBiome LLC (Industry)
Collaborators: Veristat, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MGB244-001
Record Dates: First submitted 2018-03-26; First posted 2018-04-05 (Actual); Results first posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Migraine
Keywords: Headache
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Intervention Model Description: Randomization will be 1:1:1 so that equal number of subjects will be treated in each arm of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each participant scheduled to receive investigational product (IP) will receive a randomization number at the time of randomization. The randomization number will be used to identify the study medication kit assigned to the participant and indicate the treatment to be administered to that participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- B244 Dose 1 (Experimental): B244 1X suspension in 30ml/bottle Subjects will apply 1 pump per nostril twice-a-day
  Interventions: Biological: B244
- B244 Dose 2 (Experimental): B244 4X suspension in 30ml/bottle Subjects will apply 1 pump per nostril twice-a-day
  Interventions: Biological: B244
- Vehicle (Placebo Comparator): Vehicle, 30ml/bottle Subjects will apply 1 pump per nostril twice-a-day
  Interventions: Biological: Vehicle

INTERVENTIONS:
Biological: B244 — B244 Suspension
  Arms: B244 Dose 1; B244 Dose 2
Biological: Vehicle — Vehicle Suspension
  Arms: Vehicle

SUMMARY:
This is a prospective, randomized, vehicle-controlled, double-blind, multi-center study assessing the safety, tolerability, and efficacy of B244 delivered as an intranasal spray for preventive treatment in subjects with episodic migraine.

DETAILED DESCRIPTION:
This is a Prospective, Randomized, Vehicle-controlled, Double-blind, Multi-center, 3-arm study assessing the safety, tolerability, and efficacy of B244 delivered as an intranasal spray for preventive treatment in subjects with episodic migraine.

At Screening and Baseline, all subjects must experiences 4-14 migraine days per month and 3-14 migraine attacks per month and no more than 14 headache days per month in the 3 months prior to screening.

The total duration of the study will be approximately 16 weeks. Participants will report for a Screening visit and if all inclusion criteria are met, subjects will go through a one month baseline period prior to randomization. Subjects will come in for visits at Day 28 (Week 4), Day 56 (Week8), Day 84 (Week12), and Day 112 (Week 16).

Efficacy will be assessed by change in migraine attacks, days, and hours. Blood and urine samples will be collected for standard safety laboratory testing and the effect of the drug on inflammatory biomarkers. Safety will be monitored throughout the study.

Investigators plan to enroll 303 total subjects. Subjects will be randomized 1:1:1 so that an equal number of subjects will be treated in each arm of the study.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females, 18 to 65 years of age.
* In good general health as determined by a thorough medical history and physical examination, and vital signs.
* At least a 1-year history of migraine with or without aura that began before the age of 50 years old and consistent with a diagnosis of migraine with or without aura according to the International Classification of Headache Disorders, 3rd edition, beta version.
* Experiences 4-14 migraine days per month and 3-14 migraine attacks per month and no more than 14 headache days per month (including migraine and non-migraine headache days) in the 3 months prior to screening.
* Experiences 4-14 migraine headache days per month during the baseline period.
* Ability and willingness to abstain from taking medications not allowed by the protocol or administering any foreign substance intranasally.
* Ability and willingness to complete a migraine-history diary from screening to treatment with study drug and a migraine-treatment diary from prevention treatment through the remainder of the follow-up period.

Exclusion Criteria:

* Headache on greater than 14 days/month in any of the three months (90 days) preceding entry into the study.
* Use of acute migraine-specific medications (e.g., ergotamine, triptan) on more than 10 days per month in the previous 3 months and during study.
* Use of intranasal migraine medications during study.
* Use of any intranasally administered over-the-counter product or nasal irrigation (e.g., neti pot) during study.
* Opioids/barbiturates used on more than 4 days per month in the previous 3 months and throughout the duration of the study.
* Use of analgesics (including acetaminophen, nonsteroidal anti-inflammatory drugs [NSAIDs], acetylsalicylic acid, or combination analgesics) for migraine and non-migraine headaches on more than 14 days per month in the - Use of migraine prevention medication within two months prior to study and throughout the duration of the study.
* Botulinum toxin injection within 3 months prior to screening or during study.
* Anti-CGRP monoclonal antibody (e.g., erenumab, fremanezumab, galcanezumab, and eptinezumab) injection or infusion within 4 months prior to screening or during study.
* Small molecule anti-CGRP medications in the 30 days prior to the screening visit.
* Use of systemic antibiotics during study.
* Pregnancy or breast-feeding.
* Female of childbearing potential not using adequate contraceptive measures.
* Inability to give informed consent.
* History of neurological, psychiatric, or any other medical condition that in the opinion of the investigator may compromise the subject's ability to safely participate in the study.
* Subjects with any significant clinical abnormalities which may interfere with study participation.
* Prior use of AO+ Mist.
* Subjects with immunodeficiencies, nasal lesions, nasal polyps, or sinus infections.
* Subjects who have participated in an investigational drug trial in the 30 days prior to the screening visit.
* Inability to maintain at least 80% diary compliance during the study from baseline to follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Ng-Cashin, MD, Study Director — Chief Medical Officer
Locations (22):
- United States (22):
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - CI Trials, Riverside, California
  - Neurological Research Institute, Santa Monica, California
  - New England Institute for Neurology and Headache (NEINH)/Medical Practice, Stamford, Connecticut
  - Clinical Neuroscience Solution, Inc, Jacksonville, Florida
  - Precision Clinical Research, Lauderdale Lakes, Florida
  - Clinical Neuroscience Solution, Inc, Orlando, Florida
  - Palm Beach Research, West Palm Beach, Florida
  - Neurostudies Clinical Research, Decatur, Georgia
  - BTC of New Bedford, New Bedford, Massachusetts
  - MedVadis Research, Watertown, Massachusetts
  - Altea Research Institute, Las Vegas, Nevada
  - Rochester Clinical Research INC, Rochester, New York
  - PMG Research of Wilmington, Wilmington, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Clinical Neuroscience Solution, Inc, Memphis, Tennessee
  - FutureSearch Trials of Neurology and Sleep Lab, L.P., Austin, Texas
  - FutureSearch Trials of Dallas, L.P., Dallas, Texas
  - Texas Center for Drug Development, Houston, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- B244 Dose 1: B244 1X suspension (1x10E9 cells/ml) in 30ml/bottle Subjects will apply 1 pump per nostril twice-a-day
  B244: B244 Suspension
- B244 Dose 2: B244 4X suspension (4x10E9 cells/ml) in 30ml/bottle Subjects will apply 1 pump per nostril twice-a-day
  B244: B244 Suspension
Period: Overall Study
Arm/Group | B244 Dose 1 | B244 Dose 2 | Vehicle
Started (Number of subjects treated with study drug.) | 105 | 104 | 104
Completed | 83 | 88 | 81
Not Completed | 22 | 16 | 23
Not completed — Lost to Follow-up | 7 | 6 | 7
Not completed — Withdrawal by Subject | 8 | 7 | 7
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Protocol Violation | 3 | 2 | 6
Not completed — Subject did not meet minimum number of migraines per month | 1 | 0 | 0
Not completed — Use of prohibited medication | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Subject returned for ET visit | 0 | 1 | 0
Not completed — Sponsor's decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population included all randomized subjects who received at least 1 dose of IP and had 80% ePRO diary compliance. Subjects were analyzed according to the treatment assigned by the randomization schedule.
Groups:
- Total: Total of all reporting groups
Arm/Group | B244 Dose 1 | B244 Dose 2 | Vehicle | Total
Number analyzed (Participants) | 92 | 94 | 88 | 274
Age, Customized [Count of Participants; unit: Participants]
  <30 | 16 | 12 | 16 | 44
  ≥30 | 76 | 82 | 72 | 230
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 76 | 76 | 234
  Male | 10 | 18 | 12 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 10 | 14 | 34
  Not Hispanic or Latino | 82 | 84 | 72 | 238
  Unknown or Not Reported | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 3 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 27 | 21 | 20 | 68
  White | 61 | 69 | 66 | 196
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 0 | 4
Weight [Mean (Standard Deviation); unit: kg] | 85.09 (25.835) | 93.33 (22.791) | 89.34 (25.940) | 85.85 (24.903)
Height [Mean (Standard Deviation); unit: m] | 1.66 (0.084) | 1.66 (0.111) | 1.66 (0.089) | 1.66 (0.095)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.51 (8.569) | 30.55 (9.183) | 31.99 (8.229) | 31.00 (8.675)
BMI Category [Count of Participants; unit: Participants]
  <20 kg/m^2 | 2 | 3 | 2 | 7
  20-<25 kg/m^2 | 23 | 26 | 17 | 66
  25-<30 kg/m^2 | 30 | 20 | 19 | 69
  ≥30 kg/m^2 | 37 | 45 | 50 | 132
Smoking History [Count of Participants; unit: Participants]
  Never | 73 | 66 | 62 | 201
  Former | 17 | 19 | 12 | 48
  Current | 2 | 9 | 14 | 25
Number of Migraine Days [Mean (Standard Deviation); unit: days] | 7.4 (2.86) | 7.4 (2.71) | 8.0 (3.09) | 7.6 (2.89)
Number of Migraine Attacks [Mean (Standard Deviation); unit: attacks] | 4.9 (1.88) | 5.0 (1.46) | 5.1 (1.81) | 5.0 (1.72)
Number of Acute Migraine Specific Medication Days [Mean (Standard Deviation); unit: days] | 5.5 (3.60) | 5.5 (3.22) | 6.1 (3.85) | 5.7 (3.56)
Number of Moderate and Severe Headache Days [Mean (Standard Deviation); unit: days] — Monthly Moderate and Severe Headache Days is defined as the sum of the migraine/headache days that were rated 2 (moderate pain) or 3 (severe pain) by the subject on Migraine Pain Intensity Scoring scale. These were calculated at the end of 4-week baseline period.
  days | 5.7 (2.88) | 6.2 (3.00) | 6.3 (3.07) | 6.1 (2.98)
Number of Headache Days [Mean (Standard Deviation); unit: days] | 8.3 (3.04) | 8.4 (2.88) | 9.3 (3.44) | 8.6 (3.14)
Number of Headache Hours [Mean (Standard Deviation); unit: hours] | 97.0 (68.31) | 96.4 (65.09) | 107.7 (66.68) | 100.2 (66.65)
MIDAS Score [Mean (Standard Deviation); unit: units on a scale] — The Migraine Disability Assessment (MIDAS) questionnaire was administered to study examine the relationship between the impact of migraine and quality of life where subjects scored 5 questions on a scale of 0 to 21+ (0-5=little or no disability, 6-10=mild disability, 11-20=moderate disability, 21+=severe disability). The total score ranges from 0 to 90.
  units on a scale | 30.3 (24.23) | 45.3 (50.94) | 40.1 (50.58) | 38.6 (43.98)
HIT Score [Mean (Standard Deviation); unit: units on a scale] — The Headache Impact Test-6 (HIT-6) questionnaire was administered to examine the relationship between impact of migraine and quality of life. The total score ranges from 36 to 78 where a higher score indicates a greater impact on quality of life (Class I: 36-49, Class II: 50-55, Class III: 56-59, Class IV: 60+).
  units on a scale | 63.0 (5.77) | 64.1 (4.36) | 63.9 (4.86) | 63.7 (5.03)
MSQL Score - Role Function-Restrictive [Mean (Standard Deviation); unit: units on a scale] — The Migraine Specific Quality of Life (MSQL) questionnaire was used to examine the impact of migraine on health-related quality of life across three domains: Role Function-Restrictive (7 questions) examines the degree to which performance of daily activities is limited by migraine; Role Function-Preventive (4 questions) examines the degree to which performance of daily activities is prevented by migraine; Emotional Function (3 questions) examines feelings of frustration and helplessness due to migraine. The total score for MSQL Role Restrictive ranges from 0 (less severe) to 100 (more severe).
  units on a scale | 48.1 (18.88) | 44.1 (20.17) | 45.6 (20.65) | 45.9 (19.90)
MSQL Score - Role Function-Preventive [Mean (Standard Deviation); unit: units on a scale] — The Migraine Specific Quality of Life (MSQL) questionnaire was used to examine the impact of migraine on health-related quality of life across three domains: Role Function-Restrictive (7 questions) examines the degree to which performance of daily activities is limited by migraine; Role Function-Preventive (4 questions) examines the degree to which performance of daily activities is prevented by migraine; Emotional Function (3 questions) examines feelings of frustration and helplessness due to migraine. The total score for MSQL Role Restrictive ranges from 0 (less severe) to 100 (more severe).
  units on a scale | 63.2 (21.54) | 60.3 (22.92) | 61.8 (24.13) | 61.8 (22.82)
MSQL Score - Emotional Function [Mean (Standard Deviation); unit: units on a scale] — The Migraine Specific Quality of Life (MSQL) questionnaire was used to examine the impact of migraine on health-related quality of life across three domains: Role Function-Restrictive (7 questions) examines the degree to which performance of daily activities is limited by migraine; Role Function-Preventive (4 questions) examines the degree to which performance of daily activities is prevented by migraine; Emotional Function (3 questions) examines feelings of frustration and helplessness due to migraine. The total score for MSQL Role Restrictive ranges from 0 (less severe) to 100 (more severe).
  units on a scale | 55.9 (29.73) | 50.5 (27.23) | 50.4 (27.70) | 52.3 (28.25)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Safety and tolerability endpoints will consist of all adverse events reporting during the study duration.
Time Frame: Baseline to Day 112
Population: Safety population included all subjects who received at least 1 dose of IP. Subjects were analyzed according to the IP received.
Measure: Count of Participants; unit: Participants
Arm/Group | B244 Dose 1 | B244 Dose 2 | Vehicle
Number analyzed (Participants) | 105 | 104 | 104
Participants
  At Least 1 Treatment-Related TEAE | 18 | 13 | 17
  At Least 1 Treatment-Related Grade 3 or 4 TEAE | 1 | 0 | 1
  At Least 1 Treatment-Related Serious TEAE | 0 | 0 | 0

2. Secondary Outcome: Mean Change in Monthly Migraine Days.
Description: Subjects made daily entries to include recordings of migraine frequency, duration, and severity that included information on migraine days (experiencing migraine with or without aura in a given day).
Time Frame: Baseline to Day 84
Population: Subjects from the Intent-to-Treat Population (all randomized subjects who received at least 1 dose of IP and had 80% ePRO diary compliance) that remained in the study up to Day 84 with data collected for the respective outcome measure. Subjects were analyzed according to the treatment assigned by the randomization schedule.
Measure: Mean (Standard Deviation); unit: days per month
Arm/Group | B244 Dose 1 | B244 Dose 2 | Vehicle
Number analyzed (Participants) | 65 | 68 | 65
days per month | -3.2 (4.53) | -3.0 (4.04) | -3.4 (3.77)

3. Secondary Outcome: Mean Change in Monthly Migraine Attacks.
Description: Subjects made daily entries to include recordings of migraine frequency, duration, and severity that included information on migraine attacks (an episode of any qualified migraine headache. To distinguish an attack of long duration from two attacks or to distinguish between attacks and relapses:
  A migraine attack that is interrupted by sleep, or temporarily remits, and then recurs within 48 hours (i.e., <48 hours between the start of the migraine attack to the time of the recurrence) will be considered as one attack and not two.
  -An attack treated successfully with medication but with relapse within 48 hours (i.e., <48 hours between the start of the migraine attack to the time of recurrence) will be considered as one attack.)
Time Frame: Baseline to Day 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: attacks
Arm/Group | B244 Dose 1 | B244 Dose 2 | Vehicle
Number analyzed (Participants) | 65 | 68 | 65
attacks | -2.0 (2.83) | -2.1 (2.43) | -2.0 (2.69)

4. Secondary Outcome: Proportion of Subjects Experiencing a 50%, 75%, and 100% Reduction in Monthly Migraine Days.
Description: as for outcome 2
Time Frame: Baseline to Day 112
Population: Subjects from the Intent-to-Treat Population (all randomized subjects who received at least 1 dose of IP and had 80% ePRO diary compliance) that remained in the study up to Day 112 with data collected for the respective outcome measure. Subjects were analyzed according to the treatment assigned by the randomization schedule.
Measure: Count of Participants; unit: Participants
Groups:
- B244 Dose 2: B244 4X (4x10E9 cells/ml) suspension in 30ml/bottle Subjects will apply 1 pump per nostril twice-a-day
  B244: B244 Suspension
Arm/Group | B244 Dose 1 | B244 Dose 2 | Vehicle
Number analyzed (Participants) | 65 | 68 | 65
Participants
  Week 12 : ≥50% Reduction | 31 | 36 | 32
  Week 12 : ≥75% Reduction | 20 | 17 | 17
  Week 12 : 100% Reduction | 10 | 8 | 7
  Week 16 : ≥50% Reduction: number analyzed (Participants) | 46 | 44 | 41
  Week 16 : ≥50% Reduction | 24 | 20 | 20
  Week 16 : ≥75% Reduction: number analyzed (Participants) | 46 | 44 | 41
  Week 16 : ≥75% Reduction | 12 | 7 | 12
  Week 16 : 100% Reduction: number analyzed (Participants) | 46 | 44 | 41
  Week 16 : 100% Reduction | 10 | 3 | 3

5. Secondary Outcome: Mean Change in Monthly Acute Migraine Specific Medication Days.
Description: Subjects made daily entries to include recordings of migraine frequency, duration, and severity that included use of rescue (acute migraine specific) medications and dosing administration.
Time Frame: Baseline to Day 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Groups:
- B244 Dose 1: B244 1X (1x10E9 cells/ml) suspension in 30ml/bottle Subjects will apply 1 pump per nostril twice-a-day
  B244: B244 Suspension
Arm/Group | B244 Dose 1 | B244 Dose 2 | Vehicle
Number analyzed (Participants) | 65 | 68 | 65
days | -2.0 (5.62) | -2.5 (3.70) | -2.9 (4.26)

6. Secondary Outcome: Mean Change in Monthly Headache Days.
Description: Subjects made daily entries to include recordings of migraine frequency, duration, and severity that included information on headache days (a non-migraine headache day)
Time Frame: Baseline to Day 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | B244 Dose 1 | B244 Dose 2 | Vehicle
Number analyzed (Participants) | 65 | 68 | 65
days | -3.5 (4.66) | -3.4 (3.96) | -4.2 (3.79)

7. Secondary Outcome: Mean Change From Baseline to 12 Weeks of Treatment in Disability, as Measured by the Migraine Disability Assessment (MIDAS)
Description: The Migraine Disability Assessment (MIDAS) questionnaire was administered to study examine the relationship between the impact of migraine and quality of life where subjects scored 5 questions on a scale of 0 to 21+ (0-5=little or no disability, 6-10=mild disability, 11-20=moderate disability, 21+=severe disability). The total score ranges from 0 to 90.
Time Frame: Baseline to Day 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | B244 Dose 1 | B244 Dose 2 | Vehicle
Number analyzed (Participants) | 77 | 82 | 72
score on a scale | -10.0 (24.83) | -18.0 (39.43) | -13.8 (23.82)

8. Secondary Outcome: Mean Change From Baseline to 12 Weeks of Treatment in Monthly Headache Impact Test-6 (HIT-6) Questionnaire
Description: The Headache Impact Test-6 (HIT-6) questionnaire was administered to examine the relationship between impact of migraine and quality of life. The total score ranges from 36 to 78 where a higher score indicates a greater impact on quality of life (Class I: 36-49, Class II: 50-55, Class III: 56-59, Class IV: 60+).
Time Frame: Baseline to Day 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | B244 Dose 1 | B244 Dose 2 | Vehicle
Number analyzed (Participants) | 75 | 80 | 72
score on a scale | -4.3 (6.72) | -6.2 (7.68) | -5.7 (7.54)

9. Secondary Outcome: Mean Change From Baseline to 12 Weeks of Treatment in Monthly Migraine Specific Quality of Life Questionnaire (MSQL)
Description: The Migraine Specific Quality of Life (MSQL) questionnaire was used to examine the impact of migraine on health-related quality of life across three domains: Role Function-Restrictive (7 questions) examines the degree to which performance of daily activities is limited by migraine; Role Function-Preventive (4 questions) examines the degree to which performance of daily activities is prevented by migraine; Emotional Function (3 questions) examines feelings of frustration and helplessness due to migraine. Total score for each domain ranges from 0 to 100, where a higher score indicates greater severity.
Time Frame: Baseline to Day 84
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | B244 Dose 1 | B244 Dose 2 | Vehicle
Number analyzed (Participants) | 76 | 82 | 72
score on a scale
  Role Function-Restrictive | 15.5 (18.00) | 22.7 (23.69) | 22.3 (24.53)
  Role Function-Preventive | 10.7 (16.89) | 16.1 (22.21) | 12.5 (22.04)
  Emotional Function | 11.8 (24.77) | 19.0 (27.16) | 20.2 (27.95)

10. Other Pre Specified Outcome: Mean Change in Days Where Subject Recorded Migraine Associated Symptoms: Nausea/Vomiting, Photophobia and Sonophobia.
Description: Subjects made daily entries to include recordings of migraine frequency, duration, and severity that included information on migraine associated symptoms: nausea/vomiting, photophobia and sonophobia.
Time Frame: Baseline to Day 112
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | B244 Dose 1 | B244 Dose 2 | Vehicle
Number analyzed (Participants) | 65 | 68 | 65
days
  Change from Baseline to Week 12 | -2.3 (4.68) | -2.8 (3.49) | -2.9 (3.56)
  Change from Baseline to Week 16: number analyzed (Participants) | 46 | 44 | 41
  Change from Baseline to Week 16 | -1.6 (4.61) | -2.0 (3.93) | -1.6 (4.21)

ADVERSE EVENTS:
Time Frame: Baseline to Day 112
Description: All AEs occurring after administration of the first dose of IP and on or before the final assessment were to be reported. All AEs were to be recorded irrespective of whether they were considered drug-related. AEs were to be evaluated by the Investigator at each visit for duration, intensity, and whether the event could have been associated with the IP or other causes. All SAEs were to be reported immediately by the Investigator.
Arm/Group | B244 Dose 1 | B244 Dose 2 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/104 | 0/104
Serious Adverse Events (participants affected / at risk) | 3/105 | 0/104 | 0/104
Other Adverse Events (participants affected / at risk) | 45/105 | 42/104 | 49/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B244 Dose 1 (N=105) | B244 Dose 2 (N=104) | Vehicle (N=104)
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B244 Dose 1 (N=105) | B244 Dose 2 (N=104) | Vehicle (N=104)
Upper respiratory tract infection (Infections and infestations) | 5 | 10 | 4
Nasopharyngitis (Infections and infestations) | 3 | 2 | 5
Influenza (Infections and infestations) | 3 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 2 | 1
Tooth abscess (Infections and infestations) | 1 | 2 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 2 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Tinea versicolour (Infections and infestations) | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1
Perineal infection (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 3
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Increased viscosity of upper respiratory secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Paranasal sinus hyposecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 1
Contusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 1
Blood pressure increased (Investigations) | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0
Medication residue present (Investigations) | 1 | 0 | 1
Weight increased (Investigations) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 1
Cubital tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Facial paralysis (Nervous system disorders) | 1 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 1 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 1
Ageusia (Nervous system disorders) | 0 | 0 | 1
Anosmia (Nervous system disorders) | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Sensation of foreign body (General disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Chalazion (Eye disorders) | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0
Dental implantation (Surgical and medical procedures) | 0 | 1 | 0
Sinus operation (Surgical and medical procedures) | 1 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 2
Haemorrhage (Vascular disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor shall have 45 days to review the papers. Sponsor shall have the right to require Institution/Principal Investigator, as applicable, to remove specifically identified confidential information and/or delay the proposed publication or presentation for an additional one hundred twenty (120) days to enable Sponsor to seek patent protections.

DOCUMENTS (2):
  • Study Protocol (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/63/NCT03488563/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT03488563/SAP_001.pdf